CLINICAL TRIAL: NCT06668987
Title: A Phase I/II Study to Evaluate Safety and Efficacy of the Boron Neutron Capture Therapy (BNCT) Using B10 L-BPA as Boron Carrier in Recurrent Meningioma
Brief Title: A Study of the Boron Neutron Capture Therapy (BNCT) Using B10 L-BPA in Recurrent Meningioma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heron Neutron Medical Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-08-015B
Record Dates: First submitted 2024-10-27; First posted 2024-11-01 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Meningioma; Boron Neutron Capture Therapy
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BNCT, recurrent meningioma. (Experimental): Single arm treated by BNCT only
  Interventions: Drug: B10 L-BPA Injection

INTERVENTIONS:
Drug: B10 L-BPA Injection — The investigational product is B10 L-BPA Injection, is a boron-containing compound in which 10B replaces a position on L-phenylalanine at the para position with dihydroxyboron.

SUMMARY:
This Phase I/II study, titled 'A Study to Evaluate the Safety and Efficacy of Boron Neutron Capture Therapy (BNCT) Using B10 L-BPA as a Boron Carrier in Recurrent Meningioma', aims to assess the efficacy of B10 L-BPA with BNCT in patients with recurrent meningioma. The primary objective is to evaluate the safety and efficacy of BNCT with B10 L-BPA for recurrent meningioma treatment, using the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) as the standard for assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 20 years and older.
2. Patients with recurrent intracranial meningioma confirmed by medical imaging, classified as WHO Grade 1 to 3 according to the World Health Organization grading system for meningioma, are eligible for inclusion.
3. Prior surgery, radiation therapy, radiosurgery, proton therapy, heavy ion therapy, or boron neutron capture therapy for the disease.
4. There must be a time interval ≥ 3 months between prior radiation therapy and the scheduled BNCT.
5. There must be a time interval ≥ 1 month between receipt of antitumor drugs and the scheduled BNCT.
6. Measurable disease by magnetic resonance imaging (MRI) and/or computed tomography (CT) scan and ≤ 12 cm in the longest dimension.
7. At least one measurable lesion that can be assessed by RECIST v1.1.
8. Eastern Cooperative Oncology Group (ECOG) Performance Score ≤ 2.
9. Life expectancy ≥ 3 months in the opinion of the investigator.
10. Adequate organ functions as defined below:

    Hemoglobin ≥ 8.0 g/dL. White blood cell (WBC) count ≥ 2.5 x 10^9 /L. Neutrophil count ≥ 1.0 × 10^9/L. Platelet count ≥ 50 × 10^9/L. Aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN). Alanine aminotransferase (ALT) ≤ 2.5 × ULN. Serum creatinine ≤ 1.5 × ULN Estimated glomerular filtration rate(eGFR) >=15 mL / min / 1.73m2
11. Female subjects with reproductive potential must have a negative result of serum pregnancy test at the screening visit and urine pregnancy test before the B10 L-BPA administration.
12. Female subject with childbearing potential as well as male subject with reproductive potential must agree to refrain from unprotected sex and use 2 methods of highly effective contraception with their partner (e.g. barrier contraceptives [male condom, female condom, or diaphragm plus spermicide], intrauterine device, hormonal methods [hormone shot or injection, implants, combination oral contraceptives, or patches]) for ≥ 6 months after the BNCT until the end of this study.
13. Physically and mentally capable of participating in the study and willing to adhere to study procedures.
14. Provision of signed informed consent. -

Exclusion Criteria:

1. Patients who have an effective standard treatment option available.
2. Lymphoma or other tumor type that is expected to respond to cancer chemotherapy or to a dose of conventional radiation therapy that can be safely given.
3. History of malignancy other than meningioma within 5 years (except carcinoma in situ and non-melanoma skin cancer).
4. A time interval less than 3 months from previous radiation therapy for intracranial region.
5. Patients who had radiation myelitits or radiation necrosis of the brain/brain stem.
6. A time interval less than 3 months from last brain surgery and less than 1 month from previous chemotherapy.
7. Distant metastasis outside of skull.
8. Imaging studies demonstrating tumor invasion of the carotid artery.
9. Carotid blowout syndrome with active bleeding within 6 months.
10. The investigator will evaluate the subject's condition and determine whether to perform computed tomography angiography (CTA) to assess the health of the subject's vascular system. This evaluation will confirm whether the subject is suitable to participate in the trial.

    Note: Subjects will be eligible for the study if they have undergone stent implantation and obtained consent from the investigator.
11. Active infections requiring systemic treatment.
12. Patients with severe congestive heart failure or renal failure, as well as myocardial infarction, unstable angina, or poorly controlled arrhythmia within 6 months prior to the scheduled BNCT.
13. Severe comorbidities including but not limited to poorly controlled epilepsy, poorly controlled diabetes mellitus, poorly controlled hypertension, chronic lung diseases, e.g., obstructive pneumonia, interstitial pneumonia, pulmonary fibrosis, and severe emphysema, kidney diseases, e.g., chronic renal failure, acute renal failure, phenylketonuria and nephrotic syndrome, cardiac diseases, e.g., New York Heart Association (NYHA) Functional Classification Class III or IV), phenylketonuria and/or other severe conditions in the opinion of the investigator.
14. Suspected or known hypersensitivity (including allergy) to any of the drug components or contrast media.
15. Subject with hereditary fructose intolerance.
16. With a cardiac pacemaker or an unremovable metal implant in the head and neck region that will interfere with MRI-based dose-planning or tumor response evaluation.
17. Restless subjects who are unable to lie or sit in a cast for 30-60 mins.
18. Any medical or psychiatric conditions that, in the opinion of the investigator, may interfere with optimal participation in the study or place the subject at increased risk of adverse events (AEs).
19. Concurrent systemic cancer treatments, such as chemotherapy, targeted therapy (including cetuximab or EGFR oral tyrosine kinase inhibitors), or immunotherapy.
20. History of substance or alcohol abuse within 6 months prior to the screening visit.
21. Female subject who is planning to be pregnant or lactating during the study period.
22. Subject who is considered unfit to participate in the clinical study as assessed by the investigator -

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of BNCT using B10 L-BPA in treating recurrent meningioma | 6 months
  Safety will be assessed by monitoring the frequency and severity of treatment-emergent adverse events (TEAEs), including serious adverse events and those causing permanent discontinuation of therapy as per protocol. Additionally, safety evaluations will track changes in laboratory test results, vital signs, physical examination findings, and the Eastern Cooperative Oncology Group (ECOG) performance status.
  Efficacy of BNCT with B10 L-BPA for treating recurrent meningioma will be assessed by the percentage of subjects achieving complete response (CR) and partial response (PR). Tumor response and progression will be evaluated according to RECIST 1.1 criteria, using high-resolution CT or MRI, which defines four response categories: CR, PR, stable disease (SD), and progressive disease (PD). In addition, local control will be evaluated as a separate endpoint.

SECONDARY OUTCOMES:
Progression-free survival | 6 months
  PFS is defined as the time from receiving the B10 L-BPA-based BNCT until progressive disease (PD) or death from any cause, whenever comes the first.
Overall survival | 6 months
  Overall survival is defined as the time from receiving the B10 L-BPA-based BNCT until death from any cause.
Quality of life (QoL) | 6 months
  The EORTC QLQ-C30 questionnaire assesses quality of life through functional, symptom, and global health scales, primarily using a 4-point scale (1='Not at All' to 4='Very Much') and a 7-point scale for two items, where higher scores indicate more symptoms. The QLQ-BN20, specifically designed for brain cancer patients, evaluates symptoms and limitations related to motor and communication issues, with higher scores reflecting greater severity. Together, these tools provide a comprehensive assessment of quality of life for brain cancer patients.
  To determine whether patients' quality of life improves after BNCT with B10 L-BPA, questionnaires will be administered before treatment and at 1, 3, and 6 months post-irradiation. A decrease in QLQ-C30 and QLQ-BN20 scores after irradiation will indicate improved quality of life, and the score of participants showing this improvement will be used to evaluate the benefits of BNCT with B10 L-BPA.

OTHER OUTCOMES:
The population of circulating immune cells | 6 months
  Blood samples will be collected to assess MDSCs and T cells at multiple time points: before and after BNCT. This approach aims to clarify whether the levels of circulating immune cells could serve as prognostic indicators for BNCT treatment outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hsopital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No